CLINICAL TRIAL: NCT02932228
Title: Evaluating Innovative Care Models for High-Utilizing Patients
Brief Title: Evaluation of Intensive Management Patient Aligned Care Team
Acronym: ImPACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: VA Palo Alto Health Care System (U.S. Federal Agency); Veteran Affairs Office of Patient Care Services (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PPO 13-117
Record Dates: First submitted 2016-10-06; First posted 2016-10-13 (Estimated); Results first posted 2019-05-29 (Actual); Last update posted 2019-06-12 (Actual); Status verified 2019-05

CONDITIONS: Primary Health Care; Health Care Costs

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ImPACT (Experimental): Patients in ImPACT receive intensive outpatient care from the ImPACT team. The ImPACT team augments existing PACT primary care with intensive services delivered by a multidisciplinary team (including a physician, nurse practitioner, social worker, recreational therapist, and program coordinator). ImPACT program elements include a comprehensive patient assessment, identification and tracking of patients' goals and priorities, care management for medical and social service needs, co-attendance at specialty care appointments, and coordination of care with VA and non-VA providers, including during and after hospitalization.
  Interventions: Other: ImPACT
- PACT (No Intervention): Patients in PACT receive usual VA primary care through the VA's Patient Centered Medical Home. VA primary care is delivered by PACT teamlets that comprise a primary care provider, nurse, clinical associate, and administrative associate who are supported by social work, pharmacy, and behavioral health services.

INTERVENTIONS:
Other: ImPACT — The ImPACT team offers the following services:
  * An intensive intake process, including a home visit if deemed appropriate
  * Frequent contact (in-person, telephone, or secure messaging) tailored to a patient's needs
  * After-hours access to on-call team member in order to avoid unnecessary emergency care
  * Optimization of chronic condition management using evidence-based protocols
  * Navigation of transitions between hospital and home
  * Coordination of specialty care, including contact with specialists when indicated
  * Rapid response to signs of health status deterioration or other stressful events
  * Assess patient goals, advance directives, Physician Orders for Life-Sustaining Treatment
  Arms: ImPACT

SUMMARY:
This evaluation will examine the feasibility, implementation, and effectiveness of a quality improvement intervention-Intensive Management Patient Aligned Care Team (ImPACT)-for high-risk patients.

DETAILED DESCRIPTION:
Background: VA's highest-utilizing patients generally have complicated health care needs-including complex and multiple chronic conditions, comorbid mental health conditions, and social stressors-that contribute to high rates of hospitalization, emergency services, and specialty care use. Inspired by emerging intensive primary care models for high-utilizers, VA Palo Alto launched a quality improvement program to augment existing VA primary care (provided by Patient Aligned Care Teams, PACT) with intensive care delivered by a multidisciplinary team. The Intensive management PACT (ImPACT) intervention encompasses a number of evidence-based strategies, including a comprehensive intake process, coordination of specialty care, chronic condition case management, provision of social services, rapid response to deteriorations in health, and facilitation of transitions after high-acuity events.

The ImPACT program was designated as quality improvement (non-research) by the Palo Alto VA. A retrospective evaluation using deidentified data was approved by the Stanford University IRB.

Objectives: The objectives of this evaluation are to assess ImPACT's feasibility, implementation, and effectiveness, and lay the groundwork for future larger-scale efforts and evaluations within the VA system.

Methods: We will partner with the implementation team of VA Palo Alto's ImPACT clinic to conduct a Hybrid Type 1 evaluation of the program's feasibility, implementation, and effectiveness. Specifically, the evaluation will aim to:

1. Evaluate the feasibility and implementation of the pilot ImPACT intervention. Using semi-structured interviews with ImPACT and PACT team members and leadership, we will evaluate the success of intervention delivery, including patient identification, recruitment, and retention; provision and uptake of planned services; and monitoring of patient participation and key outcomes.
2. Evaluate ImPACT's effect on utilization and costs of care. We will use a difference-in-differences approach, wherein we compare changes in VA health care costs (total, as well as inpatient, outpatient, and fee-basis) and utilization (including hospitalizations, emergency department visits, and specialty care) among ImPACT patients and high-utilizing patients who are receiving usual PACT care.
3. Examine the association between ImPACT participation and patient-centered outcomes. Using data from surveys administered in the ImPACT clinic, we will assess patient satisfaction with the ImPACT intervention and overall care, as well as changes in patient-reported outcomes, including health status, symptom burden, and function.

ELIGIBILITY:
Inclusion Criteria:

* Patient receives care from one of 14 primary care providers (MDs, NPs) who have at least three half-days of clinic per week
* Total VA healthcare costs in the top 5% for VA Palo Alto facility during the 9-month eligibility phase (10/1/11-6/30/12) AND/OR
* Risk for one-year hospitalization in November 2012 in the top 5% (using the VA's Care Assessment Need risk-prediction algorithm)

Exclusion Criteria:

* Enrollment in VA's mental health intensive case management program, home-based primary care, or palliative care programs
* Recipient of inpatient care for over half of the 9-month eligibility phase (10/1/11-6/30/12).
* Total VA healthcare costs in the lowest cost decile in the 9-month eligibility phase (10/1/11-6/30/12)
* Risk for one-year hospitalization in November 2012 in the lowest risk quartile (using the VA's Care Assessment Need risk-prediction algorithm).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 583 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2014-06-01 (Actual); Study Completion 2015-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donna M Zulman, MD MS, Principal Investigator — VA Palo Alto Health Care System, Palo Alto, CA

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zulman DM, Jenchura EC, Cohen DM, Lewis ET, Houston TK, Asch SM. How Can eHealth Technology Address Challenges Related to Multimorbidity? Perspectives from Patients with Multiple Chronic Conditions. J Gen Intern Med. 2015 Aug;30(8):1063-70. doi: 10.1007/s11606-015-3222-9. Epub 2015 Feb 18. PMID 25691239
- [Background] Zulman DM, Pal Chee C, Wagner TH, Yoon J, Cohen DM, Holmes TH, Ritchie C, Asch SM. Multimorbidity and healthcare utilisation among high-cost patients in the US Veterans Affairs Health Care System. BMJ Open. 2015 Apr 16;5(4):e007771. doi: 10.1136/bmjopen-2015-007771. PMID 25882486
- [Background] Gidwani R, Zulman D. Association Between Acute Medical Exacerbations and Consuming or Producing Web-Based Health Information: Analysis From Pew Survey Data. J Med Internet Res. 2015 Jun 23;17(6):e145. doi: 10.2196/jmir.3801. PMID 26104000
- [Background] Breland JY, Greenbaum MA, Zulman DM, Rosen CS. The effect of medical comorbidities on male and female Veterans' use of psychotherapy for PTSD. Med Care. 2015 Apr;53(4 Suppl 1):S120-7. doi: 10.1097/MLR.0000000000000284. PMID 25767965
- [Background] Hunter G, Yoon J, Blonigen DM, Asch SM, Zulman DM. Health Care Utilization Patterns Among High-Cost VA Patients With Mental Health Conditions. Psychiatr Serv. 2015 Sep;66(9):952-8. doi: 10.1176/appi.ps.201400286. Epub 2015 May 1. PMID 25930040
- [Background] Breland JY, Chee CP, Zulman DM. Racial Differences in Chronic Conditions and Sociodemographic Characteristics Among High-Utilizing Veterans. J Racial Ethn Health Disparities. 2015 Jun;2(2):167-75. doi: 10.1007/s40615-014-0060-0. Epub 2014 Nov 8. PMID 26863335
- [Background] Hummel DL, Hill C, Shaw JG, Slightam C, Zulman DM. Nurse practitioner-led intensive outpatient team: Effects on end-of-life care. The Journal for Nurse Practitioners. 2017 Mar 14; 13(5):e245-e248
- [Result] Zulman DM, Ezeji-Okoye SC, Shaw JG, Hummel DL, Holloway KS, Smither SF, Breland JY, Chardos JF, Kirsh S, Kahn JS, Asch SM. Partnered research in healthcare delivery redesign for high-need, high-cost patients: development and feasibility of an Intensive Management Patient-Aligned Care Team (ImPACT). J Gen Intern Med. 2014 Dec;29 Suppl 4(Suppl 4):861-9. doi: 10.1007/s11606-014-3022-7. PMID 25355084
- [Result] Breland JY, Asch SM, Slightam C, Wong A, Zulman DM. Key ingredients for implementing intensive outpatient programs within patient-centered medical homes: A literature review and qualitative analysis. Healthc (Amst). 2016 Mar;4(1):22-9. doi: 10.1016/j.hjdsi.2015.12.005. Epub 2015 Dec 29. PMID 27001095
- [Result] Zulman DM, Pal Chee C, Ezeji-Okoye SC, Shaw JG, Holmes TH, Kahn JS, Asch SM. Effect of an Intensive Outpatient Program to Augment Primary Care for High-Need Veterans Affairs Patients: A Randomized Clinical Trial. JAMA Intern Med. 2017 Feb 1;177(2):166-175. doi: 10.1001/jamainternmed.2016.8021. PMID 28027338
- [Result] Wu FM, Slightam CA, Wong AC, Asch SM, Zulman DM. Intensive Outpatient Program Effects on High-need Patients' Access, Continuity, Coordination, and Engagement. Med Care. 2018 Jan;56(1):19-24. doi: 10.1097/MLR.0000000000000833. PMID 29087980

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment into ImPACT completed by ImPACT staff at VAPAHCS
Period: Overall Study
Arm/Group | ImPACT | PACT
Started | 150 | 433
Completed | 140 | 405
Not Completed | 10 | 28
Not completed — Death | 8 | 23
Not completed — not eligible upon chart review | 2 | 5

BASELINE CHARACTERISTICS:
Population: death rate before starting program, age, chronic conditions, and history of homelessness
Groups:
- Total: Total of all reporting groups
Arm/Group | ImPACT | PACT | Total
Number analyzed (Participants) | 140 | 405 | 545
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 64 | 212 | 276
  >=65 years | 76 | 193 | 269
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.4 (14) | 65.7 (13) | 66.05 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 40 | 50
  Male | 130 | 365 | 495
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 140 | 405 | 545

OUTCOME MEASURES:

1. Primary Outcome: VA Health Care Costs
Description: Estimated programs effect on cost among all patients, and correspond to the change in monthly costs among patients in impact minus the change in costs for patients in PACT.
Time Frame: 17 months
Population: Program's effect on monthly person level costs
Measure: Mean (Standard Deviation); unit: US Dollars
Groups:
- PACT: Patients in PACT receive usual VA primary care through the VA's patient centered medical home.
Arm/Group | ImPACT | PACT
Number analyzed (Participants) | 140 | 405
US Dollars
  Baseline monthly costs | 6139 (2312) | 5821 (2217)
  Follow-up monthly costs | 4850 (1780) | 4618 (1741)

2. Secondary Outcome: Hospitalization
Description: Admission rates and length of stay of acute medical/surgical, acute mental health, extended medical, and extended mental health inpatient care. Outcome reported is mean(SD) number of hospital admissions using intent to treat analysis between both groups.
Time Frame: 17 months
Measure: Mean (Standard Deviation); unit: Admissions
Arm/Group | ImPACT | PACT
Number analyzed (Participants) | 140 | 405
Admissions
  Baseline | 1.3 (1.5) | 1.3 (1.5)
  Follow-up | 0.7 (1.2) | 0.7 (1.2)

3. Secondary Outcome: Emergency Department Utilization
Description: Number of Emergency Department visits
Time Frame: 17 months
Measure: Mean (Standard Deviation); unit: visits
Arm/Group | ImPACT | PACT
Number analyzed (Participants) | 140 | 405
visits
  Baseline | 3.4 (3.3) | 3.3 (3.3)
  Follow-up | 2.1 (2.9) | 2.1 (2.9)

4. Secondary Outcome: Outpatient Utilization
Description: Number of visits to primary, specialty, and mental health clinics. Number reported is mean primary care visits between ImPACT and PACT.
Time Frame: 17 months
Measure: Mean (Standard Deviation); unit: visits
Arm/Group | ImPACT | PACT
Number analyzed (Participants) | 140 | 405
visits
  Baseline | 10.9 (7.7) | 10.6 (7.8)
  Follow up | 21.8 (17.4) | 7.4 (7.5)

5. Other Pre Specified Outcome: Feasibility: Time to Enrollment
Description: To evaluate ImPACT's feasibility, we will assess time to enrollment for invited participants. Number is reported is number of participants still enrolled in ImPACT program after 9 months
Time Frame: 9 months
Population: This analysis was only conducted on the ImPACT group.
Measure: Number; unit: participants
Arm/Group | ImPACT
Number analyzed (Participants) | 140
participants | 80

6. Other Pre Specified Outcome: Feasibility: Participation
Description: We will evaluate proportion of patients who participate in ImPACT and the frequency of their contact with ImPACT team members. Outcome measure is the average number of patient-ImPACT provider in person contacts per month from 2/2013-6/2014
Time Frame: 9 months
Population: This analysis was only conducted on the ImPACT group.
Measure: Mean (Full Range); unit: encounters
Arm/Group | ImPACT
Number analyzed (Participants) | 140
encounters | 2.4 [1 to 4]

7. Other Pre Specified Outcome: Implementation Process
Description: Interviews with ImPACT team members, PACT providers, and VA facility leadership will be used to understand the ImPACT program implementation process. Outcome measure is number of participants enrolled and completed interviews.
Time Frame: 9 months
Population: This analysis was only conducted on the ImPACT group.
Measure: Count of Participants; unit: Participants
Groups:
- Providers at VAPAHCS: Clinicians and leadership at VAPAHCS impacted by implementation of the ImPACT program
Arm/Group | Providers at VAPAHCS
Number analyzed (Participants) | 15
Participants | 15

8. Other Pre Specified Outcome: Patient Satisfaction
Description: We will assess patient satisfaction with the ImPACT intervention and changes in satisfaction with overall care. The Patient Satisfaction Questionnaires ask:
  Please describe your satisfaction with ImPACT Clinical Services
  1. Medical care
  2. Social work services
  3. Recreational and community services
  4. After-hours services
  The 4 items were combined to create a mean overall satisfaction with ImPACT care score, which ranges from 1-4, 4 indicating better satisfaction with the program. The scale is measured on a 4 point scale with 1 meaning "strongly disagree" and 4 meaning "strongly agree".
Time Frame: 9 months
Population: The survey was only given to ImPACT enrollees.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ImPACT
Number analyzed (Participants) | 50
units on a scale | 3.16 (.60)

9. Other Pre Specified Outcome: Health Status (Patient-reported)
Description: We will assess patient-reported health status through a patient survey administered at time of enrollment and 4-9 months after enrollment. Outcome measure includes mean patient activation scores between baseline and follow up survey periods. Activation is measured on a scale from 0-100, with higher numbers corresponding to higher levels of patient activation.
Time Frame: up to 9 months
Population: This analysis was only conducted on the ImPACT group.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ImPACT
Number analyzed (Participants) | 51
units on a scale
  Baseline | 62.7 (17.7)
  Follow up | 66.8 (18.2)

10. Other Pre Specified Outcome: Symptom Burden (Patient-reported)
Description: We will assess changes in patient-reported symptom burden, including pain through a patient survey administered at time of enrollment and 4-9 months after enrollment. Outcome measure below is the mean number of participants who rate their "pain in the last weeks" on a 10 point scale where 0=None and 10=severe pain, a higher value indicates worse symptom burden.
Time Frame: up to 9 months
Population: The survey was only given to ImPACT enrollees.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | ImPACT
Number analyzed (Participants) | 42
Units on a scale
  Baseline | 4.6 (3.3)
  Follow up | 4.7 (3.2)

11. Other Pre Specified Outcome: Functional Status (Patient-reported)
Description: We will assess changes in patient-reported functional status through a patient survey administered at time of enrollment and 4-9 months after enrollment. The outcome measure includes percentage of patients(from 0-100%) who indicated having some difficulty, much difficulty, or inability to perform tasks due to functional limitations. A higher score indicates more functional limitations
Time Frame: 9 months
Population: The survey was only given to ImPACT enrollees.
Measure: Number; unit: percentage of participants
Arm/Group | ImPACT
Number analyzed (Participants) | 52
percentage of participants
  Baseline | 52
  Follow up | 56

ADVERSE EVENTS:
Time Frame: 17months
Description: Adverse events required to be reported to the VA R&D and local IRB committees. A review of adverse events was completed at each annual review of the projects IRB. There were no participants affected by serious adverse events.
Arm/Group | ImPACT | PACT
Serious Adverse Events (participants affected / at risk) | 0/140 | 0/405
Other Adverse Events (participants affected / at risk) | 0/140 | 0/405

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes